CLINICAL TRIAL: NCT02469545
Title: Effect of Lactobacillus Plantarum 299v Supplementation on Major Depression Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133-47818
Record Dates: First submitted 2015-05-29; First posted 2015-06-11 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2015-08

CONDITIONS: Depression; Anxiety Disorder
Keywords: depression; microbiota-gut-brain axis; Lactobacillus Plantarum 299v; probiotic
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRI and probiotic (Active Comparator): Administering antidepressant drug (SSRI - selective serotonin reuptake inhibitor: Escitalopram or Sertraline) and probiotic (Lactobacillus Plantarum 299v) to a group of patients diagnosed with depression (n=30).
  Interventions: Drug: Lactobacillus Plantarum 299v; Drug: Escitalopram; Drug: Sertraline
- SSRI and placebo of probiotic (Placebo Comparator): Administering antidepressant drug (SSRI - selective serotonin reuptake inhibitor: Escitalopram or Sertraline) and placebo of probiotic (crystalline cellulose powder) to a group of patients diagnosed with depression (n=30).
  Interventions: Drug: Crystalline cellulose powder; Drug: Escitalopram; Drug: Sertraline

INTERVENTIONS:
Drug: Lactobacillus Plantarum 299v — Administering antidepressant drug (SSRI - selective serotonin reuptake inhibitor) and probiotic - 2x1 caps. per day of Lactobacillus Plantarum 299V (10mld colony forming units in 1 caps.) for 8 weeks.
  Arms: SSRI and probiotic
Drug: Crystalline cellulose powder — Administering antidepressant drug (SSRI - selective serotonin reuptake inhibitor) and placebo of probiotic - 2x1 placebo caps. filled with micro-crystalline cellulose powder for 8 weeks.
  Arms: SSRI and placebo of probiotic
Drug: Escitalopram — 5-20mg daily
Drug: Sertraline — 50-100mg daily

SUMMARY:
The aim of the study is to determine the influence of supplementation of probiotic Lactobacillus Plantarum 299V vs. placebo of probiotic during antidepressant monotherapy with SSRI (Selective Serotonin Reuptake Inhibitor) in patients with major depression.

DETAILED DESCRIPTION:
For period of 8 weeks patient will receive probiotic Lactobacillus Plantarum 299V or its placebo as a supplementation of regular depression treatment with SSRI (Escitalopram or Sertraline). Psychometric and biochemical parameters will be monitored and evaluated. At day one, after 3 weeks (day 21) and after 8 weeks (day 56) of the study psychometric parameters will be measured such as Hamilton Depression Rating Scale, PSS-10 Scale, SCL-90 scale. At day one and after 8 weeks (day 56) of the study cognitive functions will be measured using: CVLT- California Verbal Learning Test, RFFT Ruff Figural Fluency Test, Stroop Test, Connecting Points Test (A and B), Attention and Perceptivity Test. At day one and after 8 weeks (day 56) of the study biochemical parameters will be measured such as: morning cortisol, pro and anti-inflammatory cytokines, tryptophan and its kynurenic pathway metabolites concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Unipolar depression, with at least one depressive episode, present episode since at least 2 weeks, with Hamilton Depression Scale scoring 18 and higher with BMI =18,9 - 29,9 kg/m2

Exclusion Criteria:

* Inflammatory diseases eg. rheumatoid diseases, inflammatory bowel diseases, autoimmunological diseases
* Metabolic diseases e.g. diabetes type I,II, obesity (Body Mass Index)>30 kg/m2
* Previously diagnosed other psychiatric diseases other than depression, psychoactive substances abuse, organic brain dysfunctions
* Smokers
* Patients after surgeries in last 3 months
* Oncological patients
* Patients during pregnancy or lactation
* Drugs which might influence measured parameters (e.g. lithium, antibiotics, glucocorticosteroids, antipsychotic drugs)
* Changes in routine blood biochemical parameters: morphology, electrolytes, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), creatinine, urea, C-reactive protein (CRP), thyroid-stimulating hormone (TSH).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of psychometric parameters - Change in Hamilton Depression Rating Scale from baseline at 3 weeks and 8 weeks of the study. | At day one, after 3 weeks (day 21), after 8 weeks (day 56) of the study
Evaluation of psychometric parameters - Change in Perceived Stress Scale (PSS-10) from baseline at 3 weeks and 8 weeks of the study. | At day one, after 3 weeks (day 21), after 8 weeks (day 56) of the study
Evaluation of psychometric parameters - Change in Symptom Checklist 90 Scale (SCL-90) from baseline at 3 weeks and 8 weeks of the study. | At day one, after 3 weeks (day 21), after 8 weeks (day 56) of the study

SECONDARY OUTCOMES:
Cognitive functions evaluation - California Verbal Learning Test (CVLT) | At day one, after 8 weeks (day 56) of the study
Cognitive functions evaluation - Ruff Figural Fluency Test (RFFT) | At day one, after 8 weeks (day 56) of the study
Cognitive functions evaluation - Stroop Test (A and B) | At day one, after 8 weeks (day 56) of the study
Cognitive functions evaluation - Connecting Points Test (A and B) | At day one, after 8 weeks (day 56) of the study
Cognitive functions evaluation - Attention and Perceptivity Test | At day one, after 8 weeks (day 56) of the study
Biochemical analysis - morning cortisol level | At day one, after 8 weeks (day 56) of the study
  Biochemical analysis will be based on pro-inflammatory and anti-inflammatory cytokines measurements, morning cortisol concentration, tryptophan and its kynurenic pathway metabolites measurements.
Biochemical analysis - cytokines measurements profile | At day one, after 8 weeks (day 56) of the study
Biochemical analysis - kynurenic pathway metabolites measurements profile | At day one, after 8 weeks (day 56) of the study

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Z Rudzki, MD Psychiatry Specialist, Principal Investigator — Department of Psychiatry, Medical University of Bialystok; Napoleon Waszkiewicz, MD PhD, Study Director — Psychiatry Department of Bialystok Medical University
Locations (1):
- Department of Psychiatry, Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided